CLINICAL TRIAL: NCT04862910
Title: Effects of Kinect-based Virtual Reality Training on Bone Mineral Density, Fracture Risk, Physical Performance and Quality of Life in Postmenopausal Women With Osteopenia
Brief Title: Effects of Kinect-based Virtual Reality Training in Postmenopausal Women With Osteopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/Lhr/21/1102/B Saima Riaz
Record Dates: First submitted 2021-04-23; First posted 2021-04-28 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Postmenopausal Osteopenia
Keywords: Postmenopausal Osteopenia; Bone Mineral Density; Virtual Reality; Fracture; Quality of Life
MeSH Terms: conditions — Fractures, Bone | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinect Based Virtual Reality Training (Experimental): Kinect-Based Virtual Reality Training 30 Minutes walk outdoor Routine Medication and routine diet will be continued.
  Interventions: Other: Kinect Based Virtual Reality Training
- Control Group (Other): 30 Minutes walk outdoor Regular active life style Routine diet and routine Medication
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Kinect Based Virtual Reality Training — The participant will receive the game instructions from the examiner.Protocol will be implemented 3 steps Warm Up phase Activity phase and cool down phase. The games will be played under the supervision and guidance of the therapist.Games are selected from Kinect games Kinect Sports Kinect Adventures and Your Shape Fitness Evolved. Three treatment sessions per week will be given to each participant. Total duration of each treatment session will be 45 Minutes.Participants will be instructed to walk outdoors for 30 Minutes daily. Routine Medication and routine diet will be continued.
  Arms: Kinect Based Virtual Reality Training
Other: Control Group — * They will be instructed to walk outdoors daily for 30 Minutes.
  * They will continue their daily activities with a routine diet and routine Medication
  Arms: Control Group

SUMMARY:
Osteopenia is a clinical term to define the declined Bone Mineral Density (BMD) as per the normal reference values but not low enough to meet osteoporotic diagnostic criteria. A Dual-energy x-ray absorptiometry (DXA) bone scan is used to diagnose decreased BMD. Osteopenia is, as described by the World Health Organization (WHO), a score ranging from -1 to -2.5, whereas Osteoporosis is diagnosed with values less than - 2.5. The risk of a decrease in BMD doubles as a woman goes into Menopause. The objective of this study will be to determine the effects of Kinect-based virtual reality training on BMD, fracture risk, physical function and Quality of life in postmenopausal women with Osteopenia.

This study will be a Randomized controlled trial. The study will be conducted at Riphah Rehabilitation Center, Lahore. Duration of the study will be 18 months. The sample size will be calculated after the completion of the pilot study. Initial screening of the participants will be done as per screening protocol and participants fulfilling inclusion criteria will be randomly allocated into two groups. Group A will receive Kinect based virtual reality training along with routine diet and routine Medication. Group B will be controlled with routine diet and routine Medication. Participants of both groups will be assessed at baseline for BMD, risk of fracture, all Objective and subjective parameters of Physical Performance and Quality of Life. Post-treatment assessment of Physical performance measures and Quality of life will be done after the 12th and 24th week, while BMD and fracture risk will be measured only after the 24th week. BMD will be measured by Dual-Energy X-ray Absorptiometry (DEXA) for Lumbar spine (BMD), proximal femur (BMD), T-score and Z-score. Fracture risk will be calculated by FRAX score, which estimates a fracture's probability within the next ten years. Physical Performance will be assessed by Time Up and Go Test (TUG), Functional Reach Test, Five Times Sit to Stand Test, Grip strength, Fall Efficacy Scale International, Borg revised category-ratio scale (0 to 10 scale) and Dyspnea index. Urdu Version of ECOS-16 will be used for the evaluation of health-related Quality of life (HRQOL). Data will be analyzed on SPSS-25.

DETAILED DESCRIPTION:
Osteoporosis in Pakistan is estimated at about 9.9 million people, 7.2 million of whom are women. Moreover, an estimated 40 million Pakistanis were equally distributed in Osteopenia between men and women. Osteoporosis prevalence in Pakistan is expected to increase in future years, projected at 11.3 million in 2020 and 12.9 million in 2050. in Pakistan, respectively.

International Osteoporosis Foundation surveyed the Pakistani population in 2009. The findings of this study were based on ultrasound investigations. It was found that 40 million people ranging between 45 and 70 were Osteopenic, while almost 10 million people were found to be Osteoporotic. Osteoporosis's overall prevalence was found to be 16%, while that of Osteopenia was found to be 34%.

Regular exercise involving different functions and subsystems of the human body is beneficial all life. There is ever-growing evidence that exercise prevents at least some harmful effects of Menopause, such as bone loss, increased risk of heart disease, or chronic diseases, such as diabetes.

Wii Fit effectively balances women with bone loss. The purpose of this study was to estimate the effectiveness of a Wii Fit controlled exergame compared with traditional balancing exercises, Quality of life, fear of fall and well-being in bone loss women. The Wii group or control Group comprised thirty-eight female participants aged over 65 years with a bone loss. A supervised Wii fit equilibrium training may be helpful to improve equilibrium issues among women with bone loss.

Bone consistency is greatly affected by physical activity. The following guidelines can be made for physical activity and exercise based on data derived from controlled clinical trials and meta-analyzes (randomized/nonrandomized). 1. Adolescent and prepubertal girls will benefit most from bone loading. Education is an efficient way of growing the peak bone mass of this age group and allows for the prevention of lifelong fractures. 2. Exercises with high impacts, such as jumping or skipping, or strength training paired with movement with high or irregular impacts, are the most powerful for bone.3. In order to preserve or strengthen bone, two to four short workouts (30 mins/day or less) a week for an extended period. 4. Other weight-bearing activities such as resistance training, unique positions of yoga, aerobics, low load, or walking can preserve or boost bone density in older women with risk factors that prevent them from engaging in high impact activities. 5. Additional practices that protect or increase mobility and strength often benefit, as they reduce risk of falling and thus reduce fracture risk.

High-Intensity Resistance and Impact Training (HiRIT) Improves BMD and Physical Function in Postmenopausal Women with Osteopenia and Osteoporosis. A short, controlled, twice-week HiRIT training procedure was productive and superior to previous bone enhancement programs, clinically appropriate locations, stature, functional Performance, and falls in postmenopausal women with low to high bone mass.

Effects of circuit training interventions on bone metabolism markers and bone density of older women with Osteopenia. The conclusion indicated that the circuit training intervention showed positive effects on bone metabolism markers and bone density of older women with Osteopenia, being viewed as an effective intervention program applicable to prevent and control Osteopenia Osteoporosis in line with bone density decrease.

Given the psychological findings, VR exercise has benefited mental stress reduction and HRQOL improvement. Traditional physical therapy can be seen as a repeated and lifeless activity, which also intimidates people. Physical activity (PA) health benefits have been well established in recent decades . Despite its well-known advantages, about 25% of adults and 80% of teenagers worldwide, according to the World Health Organization (WHO), are physically inactive, somewhat through a change in culture and lifestyle. In light of psychological outcomes, VR exercise showed positive impacts on relieving mental tension and improving HRQOL.

Effects of 24 weeks of aerobic dancing on the BMD, physical fitness and health-related Quality of life (HRQOL) in postmenopausal women. The results suggested that 24-week aerobic dance intervention could lower bone fracture incidence by increasing BMD and decreasing fall risk for postmenopausal women. The program adherence in the present study was 81%. Differences were statistically detected in femoral neck BMD, muscle strength and agility.

VR exercise may positively affect the conventional exercise on individual physiological, psychological and rehabilitative outcomes. However, existing studies are far from optimal in terms of consistency, quantity and samples. To confirm these positive effects, therefore, more laborious studies are needed.

Effects of virtual reality training on postmenopausal osteoporotic women. They concluded that virtual reality training has broad beneficial effects on BMD, bone mineral content and Quality of life in postmenopausal osteoporotic women, which may further reduce the risk of osteoporotic fracture. There have been few drawbacks during the whole analysis. The sample was small, and the second sample did not examine the long-term effects of this training. In future studies, the association between BMD and the Quality of life in osteoporotic women after Menopause is proposed.

A Planned, structured and repetitive exercise program is often perceived as boring and hard, thereby causing the individuals to be away from Physical Activity-related behaviours after long days of work. Instead, individuals are more interested in leisure activities, such as video games, where entertainment can be obtained while relaxing. Thus, virtual reality-based video games may trigger their interest, motivation and adherence to exercise. To the best of the researcher's knowledge, no study has investigated the effects of Kinect-based virtual reality training on BMD, fracture risk, physical function, and Quality of life in postmenopausal women with Osteopenia. Although a study has been done to check its effects on postmenopausal women with Osteoporosis; however, considering several limitations in this study, it seemed that more scientific research needs to be done to find out the facts. Asociation between BMD and Quality of life resulting from Kinect-based virtual reality training is also recommended for further research in previous literature. Therefore, the purpose of this study will be to find out the effects of Kinect-based virtual reality training on BMD, future fracture risk, physical function, and Quality of life in postmenopausal women with Osteopenia and to find out the association between BMD and Quality of life. It is hypothesized that Kinect-based virtual reality training for 24 weeks will lead to significant improvements in the outcome measures and will contribute to its role in delaying the progress of Osteopenia to Osteoporosis in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Osteopenia verified by dual-energy X-ray absorptiometry with Lumbar spine or femur T-score between -1 to -2.5 either recommended by the study investigators or verified by a physician in the past one year.
* current body mass index (BMI) < 30 kg/m2
* Patients with Normal balance and no risk of fall checked by Tandem Stance Test (TST)

Exclusion Criteria:

* Impairment of communicative and sensorial functions, Impaired Cognition, and Neurological disorders
* Cardiovascular disease or other chronic conditions that could interfere with their safety during testing or training procedures
* Pulmonary disease requiring oxygen therapy, Symptomatic orthostatic hypotension, Moderate or severe respiratory failure
* secondary osteoporosis, arthrosis or known osteoporotic fractures, neoplastic disease
* Virtual game phobia
* Games used in past six months
* Cases with epilepsy

Ages: 48 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 52 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
DUAL-ENERGY X-RAY ABSORPTIOMETRY (DXA) | 6 Months
  The most commonly used Gold standard BMD test is a densitometric technique called DXA (dual-energy X-ray absorptiometry), which can be measured in vivo and validated by many studies for BMD, T-score and Z-Score.
WHO's FRACTURE RISK ASSESSMENT TOOL (FRAX) ALGORITHM | 6 Months
  FRAX, released in 2008 by the World Health Organization, was developed and validated under the direction of Professor John Kanis with the support of many individuals and organizations, including the American Society for Bone and Mineral Research, the National Osteoporosis Foundation, the International Society for Clinical Densitometry, and the International Osteoporosis Foundation.It calculates the 10-YEAR PROBABILITY OF OSTEOPOROTIC FRACTURE using WHO's fracture Assessment calculator with age, sex, weight, height, clinical risk factors, and femoral neck BMD.

SECONDARY OUTCOMES:
TIMED UP AND GO TEST | 6 Months
  According to Shumway Cook et al., the TUG is a sensitive and specific measure of probability for older adults' falls.The Test is considered a simple and validated method used clinically to assess the patients' functional mobility. During the administration of the Test, the patient is desired to stand up from a chair. Walk for three meters, turn back, walk back and then sit down back on the chair.
FUNCTIONAL REACH TEST | 6 Months
  The Functional Reach Test is a clinical evaluation tool for dynamical balance in one easy task. In standing, the length of an outstretched arm is measured to the maximum forward extent while maintaining a fixed support base (Physiotherapy Rehabilitation of Osteoporotic Vertebral Fracture)
MODIFIED SIT AND REACH TEST | 6 Months
  The sit and reach test is a standard indicator of the lower back and hamstring muscles' flexibility. The standard sit-and-reach box is the test management tool. Wells and Dillon (1952) described this Test for the First Time and is now widely used as a general flexibility test.
FIVE TIMES SIT-TO-STAND TEST | 6 Months
  A sit-to-stand (STS) movement is considered a fundamental prerequisite for mobility and functional independence. The FTSST measures the Time taken to stand five times from a sitting position as quickly as possible. Researchers have described its use as a measure of lower limb strength, balance control, fall risk and exercise capacity.
BORG REVISED CATEGORY-RATIO SCALE (0 TO 10 SCALE) | 6 Months
  The scale allows individuals to subjectively rate their exertion level during exercise or exercise testing (American College of Sports Medicine, 2010). It is based on the category-ratio (0-10) RPE scale (BORG-CR10) developed by Borg. The RPE scale is used to measure the intensity of exercise. The RPE scale runs from 0 - 10. The numbers relate to phrases used to rate how easy or strenuous activity.
DYSPNEA INDEX | 6 Months
  A clinical measure of shortness of breath for determining exertion levels. The Baseline Dyspnea Index (BDI) measures the severity of dyspnea at the baseline (or the beginning of a clinical trial). The Transition Dyspnea Index (TDI) measures changes from this baseline (transition period) at subsequent visits.
  Levels of shortness of breath (SOB) 0=No SOB; can count to 15 (takes about 8 seconds) without taking a breath in the sequence.
  1. Mild SOB; can count to 15 but must take one short breath in the sequence.
  2. Moderate SOBneed to take 2 breaths to count to 15 in the sequence.
  3. Definite SOB; must take 3 breaths in the sequence of counting to 15.
  4. Severe SOB; unable to count or speak
DIGITAL HAND-HELD DYNAMOMETER | 6 Months
  Hand dynamometer has excellent reliability to test grip strength. It is reported as an indicator of total body strength, an objective test for physical capability, and a valid predictor of work capacity, degree of disease/injury, and rehabilitation outcomes.
QUALITY OF LIFE EVALUATION: ECOS-16 QUESTIONNAIRE | 6 Months
  ECOS-16 was developed to evaluate Quality of life in postmenopausal osteoporotic patients based on the osteoporosis specific quality of life instruments QUALEFF and OQLQ. (62)ECOS-16 contains 12 items from QUALEFFO and four items from OQLQ. The 16 items in ECOS-16 are divided into physical functioning, pain, fear of illness and psychosocial function. Five response options are offered per item with scores varying between 1 and 5 points, where 5 represents the worst QoL score. In this study, ECOS-16 will be translated first in the Urdu language, and then after its validation check, it will be used to measure Quality of life in study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil Ur Rehman, PhD, Study Chair — Riphah International University; Saima Riaz, PhD*, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Genesis Healthcare Consultants, Lahore, Punjab Province
  - Riaz, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cranney A, Jamal SA, Tsang JF, Josse RG, Leslie WD. Low bone mineral density and fracture burden in postmenopausal women. CMAJ. 2007 Sep 11;177(6):575-80. doi: 10.1503/cmaj.070234. PMID 17846439
- [Background] Karaguzel G, Holick MF. Diagnosis and treatment of osteopenia. Rev Endocr Metab Disord. 2010 Dec;11(4):237-51. doi: 10.1007/s11154-010-9154-0. PMID 21234807
- [Background] Baig L, Mansuri FA, Karim SA. Association of menopause with osteopenia and osteoporosis: results from population based study done in Karachi. J Coll Physicians Surg Pak. 2009 Apr;19(4):240-4. PMID 19356340
- [Background] Crandall CJ, Newberry SJ, Diamant A, Lim YW, Gellad WF, Booth MJ, Motala A, Shekelle PG. Comparative effectiveness of pharmacologic treatments to prevent fractures: an updated systematic review. Ann Intern Med. 2014 Nov 18;161(10):711-23. doi: 10.7326/M14-0317. PMID 25199883
- [Background] Gil-Gomez JA, Llorens R, Alcaniz M, Colomer C. Effectiveness of a Wii balance board-based system (eBaViR) for balance rehabilitation: a pilot randomized clinical trial in patients with acquired brain injury. J Neuroeng Rehabil. 2011 May 23;8:30. doi: 10.1186/1743-0003-8-30. PMID 21600066
- [Background] Mao Y, Chen P, Li L, Huang D. Virtual reality training improves balance function. Neural Regen Res. 2014 Sep 1;9(17):1628-34. doi: 10.4103/1673-5374.141795. PMID 25368651
- [Background] Da Gama A, Fallavollita P, Teichrieb V, Navab N. Motor Rehabilitation Using Kinect: A Systematic Review. Games Health J. 2015 Apr;4(2):123-35. doi: 10.1089/g4h.2014.0047. Epub 2015 Feb 6. PMID 26181806
- [Background] Parry I, Carbullido C, Kawada J, Bagley A, Sen S, Greenhalgh D, Palmieri T. Keeping up with video game technology: objective analysis of Xbox Kinect and PlayStation 3 Move for use in burn rehabilitation. Burns. 2014 Aug;40(5):852-9. doi: 10.1016/j.burns.2013.11.005. Epub 2013 Dec 2. PMID 24296065
- [Background] Morone G, Paolucci T, Luziatelli S, Iosa M, Piermattei C, Zangrando F, Paolucci S, Vulpiani MC, Saraceni VM, Baldari C, Guidetti L. Wii Fit is effective in women with bone loss condition associated with balance disorders: a randomized controlled trial. Aging Clin Exp Res. 2016 Dec;28(6):1187-1193. doi: 10.1007/s40520-016-0578-6. Epub 2016 May 6. PMID 27154875
- [Background] Troy KL, Mancuso ME, Butler TA, Johnson JE. Exercise Early and Often: Effects of Physical Activity and Exercise on Women's Bone Health. Int J Environ Res Public Health. 2018 Apr 28;15(5):878. doi: 10.3390/ijerph15050878. PMID 29710770
- [Background] Watson SL, Weeks BK, Weis LJ, Harding AT, Horan SA, Beck BR. High-Intensity Resistance and Impact Training Improves Bone Mineral Density and Physical Function in Postmenopausal Women With Osteopenia and Osteoporosis: The LIFTMOR Randomized Controlled Trial. J Bone Miner Res. 2018 Feb;33(2):211-220. doi: 10.1002/jbmr.3284. Epub 2017 Oct 4. PMID 28975661
- [Background] Kim KH, Lee HB. Effects of circuit training interventions on bone metabolism markers and bone density of old women with osteopenia. J Exerc Rehabil. 2019 Apr 26;15(2):302-307. doi: 10.12965/jer.1836640.320. eCollection 2019 Apr. PMID 31111017
- [Background] Yu PA, Hsu WH, Hsu WB, Kuo LT, Lin ZR, Shen WJ, Hsu RW. The effects of high impact exercise intervention on bone mineral density, physical fitness, and quality of life in postmenopausal women with osteopenia: A retrospective cohort study. Medicine (Baltimore). 2019 Mar;98(11):e14898. doi: 10.1097/MD.0000000000014898. PMID 30882707
- [Background] Qian J, McDonough DJ, Gao Z. The Effectiveness of Virtual Reality Exercise on Individual's Physiological, Psychological and Rehabilitative Outcomes: A Systematic Review. Int J Environ Res Public Health. 2020 Jun 10;17(11):4133. doi: 10.3390/ijerph17114133. PMID 32531906
- [Background] Toh LS, Lai PSM, Wu DB, Bell BG, Dang CPL, Low BY, Wong KT, Guglielmi G, Anderson C. A comparison of 6 osteoporosis risk assessment tools among postmenopausal women in Kuala Lumpur, Malaysia. Osteoporos Sarcopenia. 2019 Sep;5(3):87-93. doi: 10.1016/j.afos.2019.09.001. Epub 2019 Sep 11. PMID 31728426
- [Background] El Mohsen AM, El Ghaffar HE, Nassif NS, Elhafez GM. The weight-bearing exercise for better balance program improves strength and balance in osteopenia: a randomized controlled trial. J Phys Ther Sci. 2016 Sep;28(9):2576-2580. doi: 10.1589/jpts.28.2576. Epub 2016 Sep 29. PMID 27799698
- [Background] Harding AT, Weeks BK, Lambert C, Watson SL, Weis LJ, Beck BR. A Comparison of Bone-Targeted Exercise Strategies to Reduce Fracture Risk in Middle-Aged and Older Men with Osteopenia and Osteoporosis: LIFTMOR-M Semi-Randomized Controlled Trial. J Bone Miner Res. 2020 Aug;35(8):1404-1414. doi: 10.1002/jbmr.4008. Epub 2020 Mar 30. PMID 32176813
- [Background] Kaminska MS, Miller A, Rotter I, Szylinska A, Grochans E. The effectiveness of virtual reality training in reducing the risk of falls among elderly people. Clin Interv Aging. 2018 Nov 14;13:2329-2338. doi: 10.2147/CIA.S183502. eCollection 2018. PMID 30532523
- [Background] Badia X, Diez-Perez A, Lahoz R, Lizan L, Nogues X, Iborra J. The ECOS-16 questionnaire for the evaluation of health related quality of life in post-menopausal women with osteoporosis. Health Qual Life Outcomes. 2004 Aug 3;2:41. doi: 10.1186/1477-7525-2-41. PMID 15291959